CLINICAL TRIAL: NCT06388837
Title: Evaluation of the Effect of Symphysis Onlay Bone Graft, Injectable Platelet Rich Fibrin (I-PRF) and Xenograft on Horizontal Alveolar Ridge Augmentation in Esthetic Zone. A Retrospective Study
Brief Title: Effect of Symphysis Onlay Bone Graft, Injectable Platelet Rich Fibrin (I-PRF) and Xenograft on Horizontal Alveolar Ridge Augmentation in Esthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amany Ahmed Mohamed Alaraby, Lecturer of Oral Medicine, Diagnosis and Periodontology Department, Faculty of Dentistry, October 6 University, 6 October city, Egypt, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECO6U/20- 2021
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Symphysis Onlay Bone Graft; Platelet Rich Fibrin; Xenograft; Horizontal Alveolar Ridge Augmentation; Esthetic Zone
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Symphysis Onlay bone graft with injectable platelet rich fibrin placement) (Experimental): Patients underwent mandibular symphysis Onlay bone graft mixed with injectable platelet rich fibrin (I-PRF) placement.
  Interventions: Other: Injectable Platelet Rich Fibrin
- Group II (Symphysis Onlay bone graft mixed with Xenograft) (Experimental): Patients underwent mandibular symphysis Onlay bone graft mixed with Xenograft (InterOss® Anorganic Cancellous Granules).
  Interventions: Other: Xenograft

INTERVENTIONS:
Other: Injectable Platelet Rich Fibrin — Patients underwent mandibular symphysis Onlay bone graft mixed with injectable platelet rich fibrin (I-PRF) placement.
  Arms: Group I (Symphysis Onlay bone graft with injectable platelet rich fibrin placement)
Other: Xenograft — Patients underwent mandibular symphysis Onlay bone graft mixed with Xenograft (InterOss® Anorganic Cancellous Granules).
  Arms: Group II (Symphysis Onlay bone graft mixed with Xenograft)

SUMMARY:
The aim of the study: was to evaluate whether mandibular symphysis Onlay autogenous bone graft mixed with Injectable PRF could offer any advantages for patients undergoing horizontal alveolar ridge widening regarding increase alveolar ridge width compared to mandibular symphysis Onlay autogenous bone graft mixed with Xenograft

DETAILED DESCRIPTION:
Alveolar bone resorption is one of complications post-extraction complications where there is a reduction in the dimensions and quality of the alveolar bone. Alveolar bone resorption is known to occur over time, but resorption in the first few months of tooth extraction is known to be very significant.

The ideal bone graft material should have osteoconductive, osteogenic, and osteoinductive properties and mechanical stability and be free from disease. Osteoconductive is a physical property of a material that provides a framework for the growth of blood vessels and osteoprogenitor cells in bone formation. Osteoinductiveness is the ability to stimulate stem cells to differentiate in mature cells through stimulation by local growth factors. Osteogenicity is the bone growth factors in bone grafts.

Growth factors from PRF such as platelet-derived growth factor (PDGF), transforming growth factor (TGF), and insulin growth factor (IGF) are known to play a significant role in healing and bone regeneration to prevent excessive alveolar resorption after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 40 years.
* Both sexes.
* Patients suffering from horizontal alveolar ridge deficiency in anterior maxilla with labio-palatal dimensions less than 4 mm.
* Patients with adequate vertical ridge height compared to the neighboring alveolar bone.
* Patients with good oral hygiene and adjacent teeth bounding the empty span (span ranged from 1 to 4 missing teeth), should have healthy periodontium, intact or properly restored.
* Patients were apparently free from any systemic disease that may affect normal healing process of bone.

Exclusion Criteria:

* Patients suffering from any systemic diseases were excluded from the study.
* Poor oral hygiene and motivation.
* General contraindications to implant surgery.
* Uncontrolled diabetes.
* Irradiation, chemotherapy, or immunosuppressive therapy over the past 5 years.
* Active periodontitis.
* Psychiatric problems.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge width | 6 months postoperative
  Cone beam computed tomography (CBCT) was done to all patients to measure alveolar ridge width at the following intervals: pre-operative and 6 months postoperative.

SECONDARY OUTCOMES:
Bone density | 6 months postoperative
  Cone beam computed tomography (CBCT) was done to all patients to measure bone density at the following intervals: pre-operative and 6 months postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.